CLINICAL TRIAL: NCT04070404
Title: Study of Preoxygenation Quality Prior to General Anesthesia in Emergency Surgery
Brief Title: Quality of Preoxygenation in Emergency Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vilnius University (Other)
Responsible Party: Sponsor
Other Study IDs: 19BMT30
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Preoxygenation; Anaesthesia; Emergencies; Surgery
Keywords: Anaesthesia; Preoxygenation
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preoxygenation prior to general anaesthesia prolongs safe apnea time. Proper preoxygenation is always a challenge in emergency surgery.

The aim of our study is to estimate problems encountered during preoxygenation, their risk factors and ways of solving them.

DETAILED DESCRIPTION:
Factors, that are associated with compromised preoxygenation will be determined during our study. Pulse oximetry data and end-tidal oxygen concentration values will be evaluated in association with risk factors for insufficient anaesthesia face mask seal, difficult intubation, preoxygenation techniques used, comorbidities, physical status, hemodynamic and laboratory measures.

Parameters analysed:

* Preoperative: medical history, physical examination, laboratory findings, anthropometric data
* Intraoperative: preoxygenation equipment and method used (defined by anaesthesiologist in charge of the case), oxygenation and haemodynamic values recorded during preoxygenation and induction of anaesthesia, intraoperative laboratory values (if obtained)

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* patient going for emergency surgery under general anaesthesia
* age > 18 years

Exclusion Criteria:

* informed consent refusal
* noneligible for preoxygenation before general anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients undergoing general anaesthesia for emergency surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Efficient preoxygenation in preset time | 300 seconds
  End-tidal oxygen concentration values

SECONDARY OUTCOMES:
Factors influencing preoxygenation quality | 300 seconds
  Medical history, physical status, lab findings, preoxygenation equipment and method

CONTACTS AND LOCATIONS:
Locations (1):
- Vilnius University Hospital Santaros Clinics, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No